CLINICAL TRIAL: NCT00220025
Title: A Study To Determine the Efficacy of Whole Body Narrowband UVB Phototherapy in People With Darker Skin Types
Brief Title: Narrowband UVB Light Therapy to Patients With Dark Skin Types Who Have 10% of Their Body Involved With Psoriasis Vulgaris.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mary Sullivan-Whalen (Other)
Responsible Party: Sponsor-Investigator, Mary Sullivan-Whalen, Co-Investigator, Rockefeller University
Organization: Rockefeller University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JKR-0338
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — Phototherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NBUVB (Experimental)
  Interventions: Device: Phototherapy

INTERVENTIONS:
Device: Phototherapy — The patient begins total body NBUVB that day at a dose that is 50% of the MED. Patients are treated 3-7 times per week, with increasing doses at every treatment if no burning occurs. This is continued until clearance of disease or maximum efficacy.

SUMMARY:
This study offers narrowband UVB light therapy to patients with both light and dark skin types who have 10% of their body involved with psoriasis vulgaris.

DETAILED DESCRIPTION:
Two groups of patients, having 10% of their body surface area involved with psoriasis vulgaris, will receive narrowband phototherapy. One group will have skin type I-IV, or light skin and the second group will have dark skin, or type V-VI.

All patients will receive phototherapy, with narrowband UVB, three times a week for six weeks, or a total of 18 treatments. 6mm punch skin biopsies will be done prior to starting therapy and at the completion of the study. Clinical assessments and photography will be done parallel to the skin biopsies. Results (clinically and histologically) of both groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

Patients must have stable psoriasis vulgaris, which covers at least 10% of their bodies, for at least six months. Patients can not have not been treated with narrowband UVB in the past, although other light therapies are acceptable (i.e. broadband UVB and PUVA). Patients are not allowed to receive other therapies for their psoriasis, internal and topical, while they are participating in the study. Patients may continue using non-medicated moisturizer.

-

Exclusion Criteria:

-

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 1999-06; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Clinical and histological improvement of psoriasis | beginning and end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: James G. Krueger, MD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University Hospital, New York, New York, United States

REFERENCES:
- [Derived] Johnson-Huang LM, Suarez-Farinas M, Sullivan-Whalen M, Gilleaudeau P, Krueger JG, Lowes MA. Effective narrow-band UVB radiation therapy suppresses the IL-23/IL-17 axis in normalized psoriasis plaques. J Invest Dermatol. 2010 Nov;130(11):2654-63. doi: 10.1038/jid.2010.166. Epub 2010 Jun 17. PMID 20555351